CLINICAL TRIAL: NCT04292613
Title: The Effect of Hemiplegic Shoulder Pain on Balance, Upper Extremity Function and Quality of Life"
Brief Title: "The Effect of Hemiplegic Shoulder Pain on Balance, Upper Extremity Function and Quality of Life"
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Sibel Gayretli Atan, Physiotherapist, Istanbul University
Other Study IDs: ''SBU''
Record Dates: First submitted 2020-03-01; First posted 2020-03-03 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Hemiplegic Shoulder Pain
Keywords: shoulder pain, hemiplegic, function, balance
MeSH Terms: conditions — Shoulder Pain | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: "The Effect of Hemiplegic Shoulder Pain on Balance, Upper Extremity Function and Quality of Life" — The Effect of Hemiplegic Shoulder Pain on Balance, Upper Extremity Function and Quality of Life"

SUMMARY:
"The Effect of Hemiplegic Shoulder Pain on Balance, Upper Extremity Function and Quality of Life"

DETAILED DESCRIPTION:
Hemiplegic shoulder pain is a common symptom. Our aim in this study is to investigate the relationship between hemiplegic shoulder pain and balance and upper extremity functions.

ELIGIBILITY:
Inclusion Criteria:

* Having had a cerebrovascular accident
* Ages ranging from 40 to 75
* Right or left hemiplegic
* Without mental problems
* Cooperative
* According to Brunnstrom staging, upper extremity stage 1-2-3-4-5

Exclusion Criteria:

* who do not want to be evaluated
* Under the age of 40 and over the age of 75
* Non-cooperative
* Another orthopedic shoulder problem
* Newly operated patients will not be included in the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: hemiplegic shoulder pain
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-08-03 (Actual)

PRIMARY OUTCOMES:
Upper Extremite Fugl-Meyer Assessment (UA-FMA) | 1 day (Evaluation will be done once)
  Upper Extremite Fugl-Meyer Assessment (UA-FMA) is a scale that evaluates upper extremity functionality. The total score is at least 0 and at most 66 and the high scores are positively correlated with the normal function.

SECONDARY OUTCOMES:
McGill Melzack Pain Questionnaire | 1 day (Evaluation will be done once)
  McGill Melzack Pain Questionnaire is used to assess pain. High scores are positively correlated with pain.
Short Form- 36 | 1 day (Evaluation will be done once)
  SF-36 will be used to assess physical and mental health-related quality of life. The total score is at least 0 and at most 100, and the high scores are positively correlated with high quality of life.
Berg Balance Scale | 1 day (Evaluation will be done once)
  Berg balance scale is a scale used to evaluate balance.The total score is at least 0 and at most 56, and the high scores are negatively correlated with high quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Gayretli Atan, Principal Investigator — istanbul physical therapy and rehabilitation training and research hospital
Locations (1):
- Istanbul Physical Therapy and Rehabilitation Training and Research Hospital, Bahçelievler, Istanbul, Turkey (Türkiye)